CLINICAL TRIAL: NCT00943436
Title: The Effects of Exercise on Energy Balance and Macronutrient Intake in College-aged Males
Brief Title: The Effects of Exercise on Dietary Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Univ. of Tennessee IRB:7679B
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-04

CONDITIONS: Active Lifestyle Males; Inactive Lifestyle Males
Keywords: Exercise; Sedentary; Energy Expenditure; Energy Balance; Macronutrient Intake; Energy and Macronutrient intake; Exercise and Energy Balance
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active males (Active Comparator): Males who participate in at least 30 minutes of physical activity on 5 or more days per week for the last month.
  Interventions: Other: Exercise Session; Other: Rest Session
- Inactive males (Active Comparator): Males who participate in less than 1 hour of physical activity per week for the last month.
  Interventions: Other: Exercise Session; Other: Rest Session

INTERVENTIONS:
Other: Exercise Session — This study consists of two laboratory sessions. Participants will be randomly assigned to the order in which they go through these two sessions. The "Exercise Session" will consist of the participant coming into the lab and completing 45 min bout of exercise on an exercise bike, followed by a 60 min resting period, followed by the lunch buffet portion of the session where they will have 25 min to eat ad libitum.
Other: Rest Session — This study consists of two laboratory sessions. Participants will be randomly assigned to the order in which they go through these two sessions. The "Rest Session" will consist of the participant coming into the lab and completing a 45 min period of reading followed by a 60 min resting period, followed by the lunch buffet portion of the session where they will have 25 min to eat ad libitum.

SUMMARY:
The purpose of this study is to determine whether or not energy and macronutrient intake changes when comparing habitually active and habitually sedentary college-aged males in two different sessions of one resting and one exercise.

DETAILED DESCRIPTION:
Obesity is a consequence of positive energy balance, in which more energy is consumed than expended. It is hypothesized that regular amounts of physical activity may be important in helping individuals more accurately regulate energy balance. More research is needed to understand the impact of a physically active lifestyle on energy regulation capabilities Therefore, this study looks at sedentary college aged males compared to active college aged males when looking at two different sessions of energy expenditure, one exercise session and one resting session, and their energy and macronutrient intake after these sessions. The sessions will take place in the morning where each participant will exercise or rest and then be allowed to eat from a buffet ad libitum, where acute energy and macronutrient intake will be assessed.

The following hypotheses are proposed:

* Individuals who regularly engage in physical activity will more accurately respond to an energy deficit caused by an acute period of physical activity by increasing intake at a subsequent meal.
* Individuals who do not regularly engage in physical activity (sedentary individuals) will be less sensitive to accurately regulate energy balance and will not respond to an energy deficit caused by a period of acute physical activity.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 20-25
* Percent body fat of 10-18%
* Exercises greater than or equal to 5 days/wk at 30 min/day or less than or equal to 1 day/week at 1 hour/day consistently for the past month
* Likes study foods

Exclusion Criteria:

* Does not fit in exercise criteria
* Allergies or unwillingness eat study food, falls
* From survey qualifies as a "conscious eater"

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, RD, Study Chair — University of Tennessee, Knoxville
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 male students attending the University of Tennessee were recruited to participate through ads and flyers posted around campus. The recruitment period started in November 2008 and ended in August 2009 upon completion of the study. The initial phone screen conducted to determine eligibility occurred in the HEAL lab.
Pre-assignment Details: Participants were randomly assigned to which session, exercise or rest, they engaged in first. As this is a crossover design, participants did complete both the exercise and rest conditions.
Groups:
- Active Lifestyle Males: Males that exercise greater than or equal to 5 days/wk at 30 min/day
- Inactive Lifestyle Males: males that exercise less than or equal to 1 day/week at 1 hour/day
Period: Exercise Session: 45 Minutes of Activity
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Rest Session: 45 Minutes of Reading
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.40 (2.066) | 20.90 (1.792) | 21.15 (2.000)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Energy Intake at the Meal (Exercise Session)
Description: Energy intake was measured by weighing each item served in the ad libitum buffet meal before and after the subject's meal and subtracting the difference to determine gram weight of each item consumed. Food labels and the NDS-R software were used to determine dietary intake based upon gram weight of each food consumed.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: kilocalories
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Number analyzed (Participants) | 10 | 10
kilocalories | 1105.6 (389.2) | 934.8 (222.0)

2. Primary Outcome: Energy Intake at the Meal (Rest Session)
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: kilocalories
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Number analyzed (Participants) | 10 | 10
kilocalories | 1016.8 (396.7) | 1073.0 (470.3)

3. Primary Outcome: Percent Energy From Carbohydrate at the Meal (Exercise Session)
Description: Carbohydrate intake was measured by weighing each item served in the ad libitum buffet meal before and after the subject's meal and subtracting the difference to determine gram weight of each item consumed. Food labels and the NDS-R software were used to determine dietary intake based upon gram weight of each food consumed.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of kilocalorie intake
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Number analyzed (Participants) | 10 | 10
percentage of kilocalorie intake | 41.7 (2.3) | 47.67 (7.4)

4. Primary Outcome: Percent Energy From Carbohydrate at the Meal (Rest Session)
Description: as for outcome 3
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of kilocalorie intake
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Number analyzed (Participants) | 10 | 10
percentage of kilocalorie intake | 43.7 (3.1) | 46.31 (5.0)

5. Primary Outcome: Percent Energy From Protein at the Meal (Exercise Session)
Description: Protein intake was measured by weighing each item served in the ad libitum buffet meal before and after the subject's meal and subtracting the difference to determine gram weight of each item consumed. Food labels and the NDS-R software were used to determine dietary intake based upon gram weight of each food consumed.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of kilocalorie intake
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Number analyzed (Participants) | 10 | 10
percentage of kilocalorie intake | 24.5 (4.5) | 19.78 (3.7)

6. Primary Outcome: Percent Energy From Protein at the Meal (Rest Session)
Description: as for outcome 5
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of kilocalorie intake
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Number analyzed (Participants) | 10 | 10
percentage of kilocalorie intake | 23.3 (4.7) | 21.54 (3.0)

7. Primary Outcome: Percent Energy From Fat at the Meal (Exercise Session)
Description: Fat intake was measured by weighing each item served in the ad libitum buffet meal before and after the subject's meal and subtracting the difference to determine gram weight of each item consumed. Food labels and the NDS-R software were used to determine dietary intake based upon gram weight of each food consumed.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of kilocalorie intake
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Number analyzed (Participants) | 10 | 10
percentage of kilocalorie intake | 33.8 (4.3) | 32.58 (5.1)

8. Primary Outcome: Percent Energy From Fat at the Meal (Rest Session)
Description: as for outcome 7
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of kilocalorie intake
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Number analyzed (Participants) | 10 | 10
percentage of kilocalorie intake | 33.1 (3.6) | 32.16 (6.4)

ADVERSE EVENTS:
Arm/Group | Active Lifestyle Males | Inactive Lifestyle Males
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No